CLINICAL TRIAL: NCT01271790
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating 16 and 24 Weeks of Four-Drug Regimen and 24 Weeks of a Three-Drug Regimen of GS-9451, Peginterferon Alfa 2a (PEG, Pegasys®) and Ribavirin (RBV, Copegus®) With and Without Tegobuvir (GS-9190) Followed by Response Guided PEG and RBV in Treatment Naïve Subjects With Chronic Genotype 1 Hepatitis C Virus Infection (Protocol No. GS US 196 0140
Brief Title: A Study of Response-Guided Duration of Combination Therapy With GS-9451, Pegasys® and Copegus® With and Without Tegobuvir (GS-9190) in Previously Untreated Subjects With Genotype 1 Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-196-0140
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; HCV; Rapid Virologic Response; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; HCV RNA; Polymerase inhibitor; Protease inhibitor; Treatment naïve; GS-9190; GS-9451
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — tegobuvir; GS-9451; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Active Comparator): GS-9451 and Tegobuvir (GS-9190) in combination with Pegasys® and Copegus® for 16 or 24 weeks; Pegasys® and Copegus® may be continued for up to 48 weeks total duration depending on individual response to therapy
  Interventions: Drug: Tegobuvir (GS-9190); Drug: GS-9451; Biological: Pegasys®; Drug: Copegus®
- Arm 2 (Active Comparator): GS-9451 (active) and Tegobuvir (GS-9190) placebo in combination with Pegasys® and Copegus® for 24 weeks; Pegasys® and Copegus® may be continued for up to 48 weeks total duration depending on individual response to therapy
  Interventions: Drug: GS-9451; Drug: Tegobuvir placebo; Biological: Pegasys®; Drug: Copegus®
- Arm 3 (Placebo Comparator): Placebo matching Tegobuvir (GS-9190) and GS-9451 in combination with Pegasys® and Copegus® for 24 weeks; Pegasys® and Copegus® will be continued for up to 48 weeks total duration
  Interventions: Drug: Tegobuvir placebo; Drug: GS-9451 placebo; Biological: Pegasys®; Drug: Copegus®

INTERVENTIONS:
Drug: Tegobuvir (GS-9190) — Tegobuvir (GS-9190) capsule, 30 mg BID
  Arms: Arm 1
Drug: GS-9451 — GS-9451 tablet, 200 mg once daily (QD)
  Arms: Arm 1
Biological: Pegasys® — peginterferon alfa-2a (solution for injection) 180 µg/week
  Arms: Arm 1
Drug: Copegus® — ribavirin tablet (weight based: 1000 mg/day <75 kg; 1200 mg/day ≥ 75 kg) divided twice daily (BID)
  Arms: Arm 1
Drug: GS-9451 — GS-9451 tablet, 200 mg QD
  Arms: Arm 2
Drug: Tegobuvir placebo — placebo matching Tegobuvir (GS-9190) capsule BID
  Arms: Arm 2
Biological: Pegasys® — peginterferon alfa-2a (solution for injection) 180 µg/week
  Arms: Arm 2
Drug: Copegus® — ribavirin tablet (weight based: 1000 mg/day <75 kg; 1200 mg/day ≥ 75 kg) divided twice daily (BID)
  Arms: Arm 2
Drug: Tegobuvir placebo — placebo matching Tegobuvir (GS-9190) capsule BID
  Arms: Arm 3
Drug: GS-9451 placebo — placebo matching GS-9451 tablet QD
  Arms: Arm 3
Biological: Pegasys® — peginterferon alfa-2a (solution for injection) 180 µg/week
  Arms: Arm 3
Drug: Copegus® — ribavirin tablet (weight based: 1000 mg/day <75 kg; 1200 mg/day ≥ 75 kg) divided twice daily (BID); tablet
  Arms: Arm 3

SUMMARY:
This phase 2b study will evaluate the efficacy and safety of 16 and 24 weeks of a 4-drug regimen with GS-9451 and Tegobuvir and 24 weeks of a 3-drug regimen of GS-9451 without Tegobuvir, all with Peginterferon Alfa-2a (Pegasys®) and Ribavirin (Copegus®).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 18 to 70 years of age
* Chronic HCV infection for at least 6 months prior to Baseline (Day 1)
* Liver biopsy results (performed no more than 2 years prior to Screening) indicating the absence of cirrhosis
* Monoinfection with HCV genotype 1a or 1b
* HCV treatment-naïve
* Body mass index (BMI) between 18 and 36 kg/m2
* Creatinine clearance ≥ 50 mL/min
* Subject agrees to use highly effective contraception methods if female of childbearing potential or sexually active male.
* Screening laboratory values within defined thresholds for alanine aminotransferase (ALT), aspartate aminotransferase (AST), leukopenia, neutropenia, anemia, thrombocytopenia, thyroid stimulating hormone (TSH), potassium, magnesium

Exclusion Criteria:

* Autoimmune disease
* Decompensated liver disease or cirrhosis
* Poorly controlled diabetes mellitus
* Severe psychiatric illness
* Severe chronic obstructive pulmonary disease (COPD)
* Serological evidence of co-infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or another HCV genotype
* Suspicion of hepatocellular carcinoma or other malignancy (with exception of certain skin cancers)
* History of hemoglobinopathy
* Known retinal disease
* Subjects who are immunosuppressed
* Subjects with known, current use of amphetamines, cocaine, opiates (i.e., morphine, heroin), methadone, or ongoing alcohol abuse
* Subjects who are on or are expected to be on a potent cytochrome P450 (CYP) 3A4 or Pgp inhibitor, or a QT prolonging medication within 2 weeks of Baseline (Day 1) or during the study
* Subjects must have no history of clinically significant cardiac disease, including a family history of Long QT syndrome, and no relevant electrocardiogram (ECG) abnormalities at screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response | 24 weeks of off-treatment follow-up
  Sustained virologic response (SVR) defined as undetectable hepatitis C virus (HCV) RNA 24 weeks after treatment cessation

SECONDARY OUTCOMES:
Safety and tolerability of therapy | Through treatment period and 24 weeks of off-treatment follow-up
  Safety and tolerability of therapy as measured by frequency of laboratory abnormalities, reported adverse events, and discontinuations due to adverse events
Emergence of viral resistance following initiation of therapy with GS 9190 and GS 9451 | Through treatment period, 24 weeks of off-treatment follow-up, and up to 48 weeks of follow-up in the Resistance Registry Substudy
Viral dynamics and steady state pharmacokinetics | Through Week 4 of therapy
  Viral dynamics and steady state pharmacokinetics of GS 9190 and GS 9451 when administered in combination with PEG and RBV; measured by HCV RNA levels and plasma concentrations of GS-9190 and GS-9451 over time
Durability of response in subjects who achieve SVR | 36 months following Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Bittoo Kanwar, Study Director — Gilead Sciences
Locations (144):
- United States (85):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Alabama Liver and Digestive Specialists, Montgomery, Alabama
  - Mayo Clinic, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Pacific Oaks Medical Group, Beverly Hills, California
  - eStudySite, Chula Vista, California
  - Scripps Clinic, La Jolla, California
  - eStudySite, La Mesa, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Synergy Clinical Research Center, National City, California
  - eStudySite, Oceanside, California
  - RESEARCH and EDUCATION, INC, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - Kaiser Permanente, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - South Denver Gastroenterology, Englewood, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Bach and Godofsky Infectious Diseases, Bradenton, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - University of Florida, Gainesville, Florida
  - Palmetto Research, Hialeah, Florida
  - University of Miami, Miami, Florida
  - Scientific Clinical Research, Inc c/o Segal Institute for Clinical Research, North Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Florida Hospital, Orlando, Florida
  - South Florida Center of Gastroenterology, LLC, Wellington, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Emory University, Infectious Disease Clinic, Atlanta, Georgia
  - Liver Center of Atlanta, Atlanta, Georgia
  - Dekalb Gastroenterology, Decatur, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - IGRF, Indianapolis, Indiana
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Digestive Disease Associates, PA, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Partners in Internal Medicine, P.C., Worcester, Massachusetts
  - Henry Ford Health System-Columbus center, Novi, Michigan
  - MN Gastroenterology, P.A., Plymouth, Minnesota
  - Gastrointestinal Associates, PA, Jackson, Mississippi
  - Digestive Health Specialists, PA, Tupelo, Mississippi
  - Saint Louis University, St Louis, Missouri
  - Comprehensive Clinical Research, Berlin, New Jersey
  - ID Care 105, Hillsborough, New Jersey
  - Atlantic Research Affiliates, LLC, Morristown, New Jersey
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - UNM Health Sciences Center, Albuquerque, New Mexico
  - Binghamton Gastroenterology, Binghamton, New York
  - North Shore University Hospital, Manhasset, New York
  - Concorde Medical Group, New York, New York
  - NYU Hepatology Associates, New York, New York
  - Cornell University Gastroenterology & Hepatology, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Consultants for Clinical, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - James H. Quillen VA Medical Center, Mountain Home, Tennessee
  - Columbia Medical Group, The Frist Clinic, Nashville, Tennessee
  - The North Texas Research Institute, Arlington, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Kelsey Research Foundation, Houston, Texas
  - Advanced Liver Therapies, Houston, Texas
  - Research Specialists of Texas, Houston, Texas
  - Amcare Research Inc., Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia
  - Liver Institute of Virginia, Bon Secours, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Virginia Mason Medical Center, Digestive Disease Institute, Seattle, Washington
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
- Austria (6):
  - Landeskrankenhaus Graz West, Graz
  - Medizinische Universität Graz, Graz
  - LKH Innsbruck, Innsbruck
  - Krankenhaus der Elisabethinen Linz GmbH, Linz
  - AKH der Stadt Wien, Vienna
  - Wilhelminenspital der Stadt Wien, Vienna
- Belgium (5):
  - Ziekenhuis Netwerk Antwerpen, Antwerp
  - ULB Erasme, Brussels
  - UCL Saint Luc, Brussels
  - UZ Antwerp, Edegem
  - Centre Hospitalier Universitaire Sart Tilman Liège, Liège
- France (10):
  - Beaujon Hospital, Clichy
  - Henri Mondor Hospital, Créteil
  - Hôpital de la Croix Rousse, Lyon
  - Saint Joseph Hospital, Marseille
  - Hôpital de I´Archet 2, Service Hépatologie, Nice
  - Centre Hospitalier Régional d'Orléans, Hôpital de la Source, Orléans
  - Hôpital Cochin, Paris
  - Groupe Hospitalier du Haut Leveque, Pessac
  - Centre Hospitalier Universitaire de Strasbourg - Hôpital Civil, Strasbourg
  - Nancy University Hospital Center, Vandœuvre-lès-Nancy
- Germany (11):
  - Charite University Medicine, Berlin
  - Leber- und Studienzentrum am Checkpoint, Berlin
  - University Hospital Bonn, Bonn
  - University Hospital Essen, Essen
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt/M
  - University Hospital Freiburg, Freiburg im Breisgau
  - Asklepios Klinik Sankt Georg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - University hospital Heidelberg, Heidelberg
  - University Hospital Leipzig, Leipzig
  - Johannes Gutenberg University Hospital, Mainz
- Netherlands (4):
  - Academisch Medisch Centrum Universiteit Van Amsterdam, Amsterdam
  - Radaboud University Nijmegen Medical Centre (UMC St Radboud), Nijmegen
  - Erasmus University Medical Center Rotterdam, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (12):
  - Wojewodzki Szpital Specjalistyczny im. K. Dluskiego Oddzial Obserwacyjno-Zakazny, Bialystok
  - Wojewodzki Szpital Obserwacyjno-Zakazny im. Tadeusza Browicza Oddział Obserwacyjno-Zakazny, Bydgoszcz
  - Szpital Specjalistyczny w Chorzowie, Chorzów
  - Niepubliczny Zakład Opieki Zdrowotnej "Pol-SaNa-Med" Sp. z o.o., Czeladź
  - Wojewodzki Szpital Zespolony w Kielcach, Kielce
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow
  - Wojewodzki Specjalistyczny Szpital im. Dr Wl. Bieganskiego w Lodzi, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
  - Radomski Szpital Specjalistyczny im. Dr Tytusa Chalubinskiego Oddzial obserwacyjno-zakazny z odcinkiem jednego dnia leczenia chorob watroby, Radom
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Wojewodzki Szpital Zakazny Oddzial Dzienny, Warsaw
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administracji w Warszawie, Warsaw
  - Wojewódzki Szpital Specjalistyczny im. J. Gromkowskiego, Wroclaw
- United Kingdom (11):
  - Queen Elizabeth Hospital, Birmingham
  - Royal Liverpool University Hospital, Liverpool
  - Barts and The London Hospital, London
  - Royal Free Hospital, London
  - Kings College Hospital, London
  - Chelsea and Westminster Hospital, London
  - Saint Mary's Hosptial, London
  - Manchester Royal Infirmary, Manchester
  - North Manchester General Hospital, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Derriford Hospital, Plymouth